CLINICAL TRIAL: NCT06388889
Title: An Open-Label Long-Term Phase III Extension Study to Assess the Long-Term Safety and Tolerability of Dexpramipexole in Participants With Severe Eosinophilic Asthma
Brief Title: Phase III Long-Term Extension Study With Dexpramipexole
Acronym: EXHALE-5
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Program stopped due to the benefit risk profile no longer supports further development in the intended patient population.
Sponsor: Areteia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR-DEX-22-04
Record Dates: First submitted 2024-03-27; First posted 2024-04-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Eosinophilic Asthma
Keywords: Exacerbations; Severe Asthma; EXHALE-2; EXHALE-3; EXHALE-4; Uncontrolled Asthma; Asthma Attack
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 150 mg BID (Experimental): Dexpramipexole 150 mg oral tablet taken twice a day.
  Interventions: Drug: Dexpramipexole Dihydrochloride

INTERVENTIONS:
Drug: Dexpramipexole Dihydrochloride — Oral administration of dexpramipexole tablet

SUMMARY:
The goal of this clinical trial] is to evaluate the long term safety of dexpramipexole treatment in participants with severe asthma, aged ≥18 years, on Global Initiative for Asthma (GINA) 2021 [GINA, 2021] Step 4 or 5 therapy and who completed either of the Phase III studies EXHALE-2 or EXHALE-3.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who completed the double-blind study intervention treatment period during either of the Phase III studies EXHALE-2 or EXHALE-3.
2. Participants capable of giving signed informed consent/assent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
3. Negative urine pregnancy test for women of childbearing potential (WOCBP; after menarche) at the Baseline Visit/Day 1.
4. WOCBP (after menarche) must use either of the following methods of birth control, from the Baseline Visit/Day 1 through the End of Study Visit:

   1. A highly effective form of birth control (confirmed by the investigator). Highly effective forms of birth control include: true sexual abstinence, a vasectomized sexual partner, Implanon, female sterilization by tubal occlusion, any effective intrauterine device (IUD), IUD/intrauterine system, levonorgestrel intrauterine system, or oral contraceptive. -OR-
   2. Two protocol acceptable methods of contraception in tandem. Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for ≥12 months prior to the planned date of the Baseline Visit/Day 1 without an alternative medical cause. The following age specific requirements apply:
   3. Women <50 years old will be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone levels in the postmenopausal range.
   4. Women ≥50 years old will be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.

Exclusion Criteria:

1. Clinically significant change in health status during either of the Phase III studies EXHALE-2 or EXHALE-3 which in the opinion of the investigator would make the participant unsuitable for participation in this study.
2. Participants with allergy/intolerance to dexpramipexole or any of its excipients.
3. Participants who met permanent discontinuation criteria or permanently discontinued study treatment for any reason in either of the Phase III studies EXHALE-2 or EXHALE-3..
4. Treatment with selected drugs known to have a substantial risk of neutropenia in the past 30 days.
5. Pregnant or breastfeeding women.
6. Males who are unwilling to use an acceptable method of birth control during the entire study period (ie, condom with spermicide).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Number and Percentage of Participants with a Treatment Emergent Adverse Event | 52 weeks
  Summary of participants from the safety population who experienced an adverse event.
Number and Percentage of Participants with Potentially Clinically Significant Postbaseline Changes in Clinical Laboratory Evaluations | 52 weeks
  Summary of participants from the safety population who experienced potentially clinically significant postbaseline changes in hematology and chemistry results.
Number and Percentage of Participants with Potentially Clinically Significant Postbaseline Changes in Vital Signs and Body Weight | 52 weeks
  Summary of participants from the safety population who experienced potentially clinically significant postbaseline changes in vital signs (blood pressure, pulse rate, respiratory rate, and temperature) or body weight.
Number and Percentage of Participants with Potentially Significant Postbaseline Changes in Electrocardiogram Parameters | 52 weeks
  Summary of participants from the safety population who experienced potentially significant postbaseline changes in electrocardiogram parameters: heart rate, PR, QRS and QTcF intervals.

SECONDARY OUTCOMES:
Severe Asthma Exacerbations | Averaged across 52 weeks
  Annualized rate of severe asthma exacerbations over 52 weeks
Change in Asthma Control Questionnaire-6 (ACQ-6) | Day 1 (baseline), Weeks 16, 32, and 52
  ACQ-6 is simple questionnaire to measure the adequacy of asthma control and change in asthma control which occurs either spontaneously or as a result of treatment. The 6-point self-administered scale has items measuring asthma symptoms and rescue inhaler use. The ACQ score is the mean of the questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled).
Change in absolute eosinophil counts (AEC) | Day 1 (baseline), Weeks 16, 32, and 52
  Change from baseline, at Weeks 16, 32, and 52.

CONTACTS AND LOCATIONS:
Overall Officials: Sady Alpizar, MD, Principal Investigator — Clinical Research Trials of Florida, Inc.
Locations (102):
- United States (22):
  - Research Site 20001-374, Bakersfield, California
  - Research Site 20001-376, Northridge, California
  - Research Site 20001-029, Coral Gables, Florida
  - Research Site 20001-014, Greenacres City, Florida
  - Research Site 30001-291, Jacksonville, Florida
  - Research Site 20001-066, Miami, Florida
  - Research Site 20001-001, Miami, Florida
  - Research Site 20001-311, Miami, Florida
  - Research Site 20001-026, Miami, Florida
  - Research Site 30001-082, Miami, Florida
  - Research Site 20001-024, Miami, Florida
  - Research Site 20054-024, Miami, Florida
  - Research Site 30001-429, Plantation, Florida
  - Research Site 20001-004, Tampa, Florida
  - Research Site 20001-036, Elwood, Indiana
  - Research Site 20001-044, Evansville, Indiana
  - Research Site 20001-006, Flint, Michigan
  - Research Site 20001-046, St Louis, Missouri
  - Research Site 20001-355, Toms River, New Jersey
  - Research Site 20001-047, Hawthorne, New York
  - Research Site 20001-063, Toledo, Ohio
  - Research Site 30001-297, Pearland, Texas
- Argentina (14):
  - Research Site 30054-044, Buenos Aires
  - Research Site 20054-017, Buenos Aires
  - Research Site 20054-015, Buenos Aires
  - Research Site 20054-022, Buenos Aires
  - Research Site 20054-024, Buenos Aires
  - Research Site 20054-008, Buenos Aires
  - Research Site 20054-005, Córdoba
  - Research Site 30054-047, Mendoza
  - Research Site 20054-019, Mendoza
  - Research Site 20054-016, Mendoza
  - Research Site 20054-010, Mendoza
  - Research Site 20054-002, San Miguel de Tucumán
  - Research Site 20054-020, San Miguel de Tucumán
  - Research Site 20054-013, Santa Fe
- Brazil (7):
  - Research Site 20055-007, Blumenau
  - Research Site 20055-004, Porto Alegre
  - Research Site 20055-010, Porto Alegre
  - Research Site 20055-001, São Bernardo
  - Research Site 20055-003, São Paulo
  - Research Site 20055-008, São Paulo
  - Research Site 20055-002, Sorocaba
- Bulgaria (6):
  - Research Site 20359-016, Dimitrovgrad
  - Research Site 20359-008, Montana
  - Research Site 20359-010, Pernik
  - Research Site 20359-005, Rousse
  - Research Site 20359-009, Sliven
  - Research Site 20359-016, Vidin
- Georgia (7):
  - Research Site 20995-001, Kutaisi
  - Research Site 20995-005, Tbilisi
  - Research Site 20995-006, Tbilisi
  - Research Site 20995-002, Tbilisi
  - Research Site 20995-003, Tbilisi
  - Research Site 20995-004, Tbilisi
  - Research Site 20995-009, Tbilisi
- Research Site 20081-023, Tokyo, Japan
- Mexico (3):
  - Research Site 20052-002, Guadalajara
  - Research Site 20052-012, San Juan del Río
  - Research Site 20052-014, Tijuana
- North Macedonia (2):
  - Research Site 20389-004, Skopje
  - Research Site 20389-007, Skopje
- Poland (10):
  - Research Site 20048-018, Bialystok
  - Research Site 20048-006, Giżycko
  - Research Site 20048-008, Krakow
  - Research Site 20048-027, Krakow
  - Research Site 20048-033, Krakow
  - Research Site 20048-005, Lodz
  - Research Site 20048-031, Ostrów Wielkopolski
  - Research Site 20048-010, Piaseczno
  - Research Site 20048-028, Poznan
  - Research Site 20048-016, Poznan
- Romania (2):
  - Research Site 20040-002, Brasov
  - Research Site 20040-004, Brasov
- Serbia (4):
  - Research Site 20381-002, Belgrade
  - Research Site 20381-005, Belgrade
  - Research Site 20381-007, Belgrade
  - Research Site 20381-003, Valjevo
- South Africa (6):
  - Research Site 30027-010, Durban, Kwa-ZuIu Natal
  - Research Site 30027-008, Durban, KwaZulu-Natal
  - Research Site 30027-009, Cape Town, Western Cape
  - Research Site 30027-005, Durban
  - Research Site 30027-014, Durban
  - Research Site 30027-010, Durban
- South Korea (4):
  - Research Site 20082-003, Anyang-si
  - Research Site 20082-009, Daegu
  - Research Site 20082-006, Jeonju
  - Research Site 20082-008, Seoul
- Ukraine (12):
  - Research Site 20380-002, Chernivtsi
  - Research Site 20380-014, Ivano-Frankivsk
  - Research Site 20380-004, Ivano-Frankivsk
  - Research Site 20380-018, Kyiv
  - Research Site 20380-007, Kyiv
  - Research Site 20380-010, Kyiv
  - Research Site 20380-012, Kyiv
  - Research Site 20380-013, Kyiv
  - Research Site 20380-001, Ternopil
  - Research Site 20380-003, Vinnytsia
  - Research Site 20380-003, Zhytomyr
  - Research Site 20380-005, Zhytomyr
- United Kingdom (2):
  - Research Site 20044-020, Manchester
  - Research Site 20044-026, Rochdale

IPD SHARING:
Plan to Share IPD: No